CLINICAL TRIAL: NCT06154772
Title: The Effect of Color Therapy on Quality of Life, Anxiety and Fatigue Levels of Parkison Patients
Brief Title: Quality of Life, Anxiety and Fatigue Level of Parkison's Patients With Color Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 27/09/2023
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Parkinson
Keywords: Color therapy
MeSH Terms: interventions — Color Therapy

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Color Therapy (Experimental): Balancing body chakras with colors. Colors are applied to the body's chakras for 10-15 minutes.
  Interventions: Other: Color Therapy
- Control Group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Color Therapy — Color therapy will be applied to the body chakras for 10-15 minutes with colored fabrics, color therapy with water and colored light lamp.
  Arms: Color Therapy

SUMMARY:
The aim of this study was to investigate the effect of color therapy on quality of life, anxiety and fatigue levels in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Color Therapy aims to balance and heal our body's energy centers using the seven color spectrum, which helps to promote our body's own healing process. Thus good health and well-being is achieved through the balance of all these energies. Color therapy basically consists of color and character analysis with name, color therapy with chakras, programming of the pendulum, chakras and color application, color application with water, color application with colored light device.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Parkinson's disease for at least 6 months,
* Those who have not taken sleeping pills or sedative drugs,
* Not having undergone brain stimulation surgery,
* Do not have a physical illness or cognitive disability that would prevent them from understanding the education provided, and do not have a diagnosis of a psychiatric disease,
* According to the Parkinson's Fatigue Scale, the scale score is >8
* The patient or someone living in the same house with the patient is literate,
* Patients have no vision problems.

Exclusion Criteria:

* Parkinson patients who did not agree to participate in the research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life Scale (SF36) | At the end of Color Therapy (therapy 9 times in total in 3 months)
  It was developed to measure the quality of life in people with physical diseases. It is measured in 8 dimensions and 36 items: physical function, physical role difficulty, emotional role difficulty, viability, mental health, social functionality, pain, and general health perception.
Beck Anxiety Inventory (BAI) | At the end of Color Therapy (therapy 9 times in total in 3 months)
  It consists of 21 questions and a minimum score of 0 and a maximum score of 3 is obtained from each question. As a result of the answers to all questions, all answers are summed up and a total score is obtained. In the evaluation phase, the presence and level of depression is interpreted in line with the meanings expressed by the score ranges. In the evaluation, 0-9 point range defines the presence of minimal depressive symptoms, 10-16 point range defines the presence of mild depressive symptoms, 17-29 point range defines the presence of moderate depressive symptoms and 30-63 point range defines the presence of severe depressive symptoms. A score of 17 and above indicates a level of depression that may require treatment.
Parkinson's Fatigue Scale (PYO-16) | At the end of Color Therapy (therapy 9 times in total in 3 months)
  It consists of 16 items, with 5 responses for each item (1=strongly disagree, 5=strongly agree). The result evaluation can be done in two different ways. The total value is calculated as the average of the response to all items (value range 1-5). Scores above the average "3.3" are considered tired. In the other rating option, 0 (actual response 1-3) and 1 (actual response 4-5) are scored, with a total value between 0-16. A total of 8 points and above is considered tired. In both methods, a higher value indicates a higher level of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No